CLINICAL TRIAL: NCT05876416
Title: Decoding the Genetic Landscape of Skeletal Diseases
Acronym: SKDLAND
Status: Recruiting | Type: Observational
Sponsor: Karolinska Institutet (Other)
Collaborators: Karolinska University Hospital (Other); Göteborg University (Other)
Responsible Party: Principal Investigator, Giedre Grigelioniene, Associate Professor, MD, PhD, Karolinska Institutet
Other Study IDs: 910715; 2022-02647 (Other Grant/Funding Number: Vetenskap Rådet/SRC)
Record Dates: First submitted 2023-04-16; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Genetic Skeletal Diseases; Skeletal Dysplasia; Molecular Causes; Skeletal Disorder
MeSH Terms: conditions — Mucopolysaccharidosis IV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Genomic DNA samples, primary dermal fibroblasts, RNA from blood or fibroblasts
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This 5-year project aims to (1) search for genetic causes for yet unsolved congenital skeletal disorders (GSDs); (2) study consequences of the newly identified pathogenic variants in cells and in transgenic mice, (3) summarize data on natural course and complications for different GSD groups. For patients with unsolved GSD, the investigators search for molecular causes of GSDs using whole genome sequencing (WGS) and total ribonucleic acid (RNA) sequencing. Candidate gene variants are selected using genome or transcriptome sequencing data, clinical findings and screening of omics databases. Causality of the new variants is studied in cells and in transgenic mice models. Molecular and clinical findings are summarized for different GSD groups.

DETAILED DESCRIPTION:
Genetic skeletal disorders (GSDs) are a large group of rare diseases caused by abnormalities in genes regulating skeletal development. This 5-year project aims to (1) search for genetic causes for yet unsolved congenital skeletal disorders; (2) study consequences of the newly identified pathogenic variants in cells and in transgenic mice, (3) summarize data on natural course and complications for different GSD groups. The project is a collaboration between the Dept of Clinical Genetics, Karolinska University Hospital, Lab of Clinical Genetics and Lab of Bone and Cartilage Physiology, Karolinska Institutet and Sahlgrenska Academy. In a well-characterized group of 300 GSD participants whose DNA samples were analyzed using whole genome sequencing (WGS), there are 120 study participants with unsolved diagnoses. For those participants, we search for molecular causes of GSDs using WGS and total RNA sequencing. Candidate gene variants are selected using genome or transcriptome sequencing data, clinical findings and screening of omics databases. Causality of the new variants is studied in cells and in transgenic mice models. Molecular and clinical findings are summarized for different GSD groups. Our results improve diagnostics for GSDs, advance knowledge on pathogenesis and help establishing new individual follow-up and treatment strategies for patients with GSDs. This project increases understanding of skeletal pathophysiology and will contribute to the development of novel treatment methods for skeletal diseases.

ELIGIBILITY:
Inclusion Criteria:

Clinically suspected skeletal dysplasia based on previous investigations

Abnormal height

Radiographic abnormalities of the skeleton in addition to other syndromic features

Healthy relatives of the affected study participants

Exclusion Criteria:

No radiographic data available from clinical investigations

Suspected environmental or multifactorial causes

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals of any age with congenital skeletal diseases and their healthy relatives
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
New gene discoveries for genetic skeletal disorders (GSDs) | 2023-2028
  2-3 new disease causes and disease entities identified and reported per year for GSDs.
Improved knowledge regarding natural cause of rare GSDs | 2023-2028
  1-2 GSDs reported as small patient groups with the same condition and clinical characteristics/course.

SECONDARY OUTCOMES:
Disease (GSD) associated traits and complications | 2023-2028
  The observations include internal malformations, metabolic, biochemical and growth parameters, and secondary complications.
Information on disease causing variants in GSD | 2023-2028
  During the study we identify several novel disease causing variants in known GSD genes and report them to databases.

CONTACTS AND LOCATIONS:
Overall Officials: Giedre Grigelioniene, MD,, Principal Investigator — Dept Molecular Medicine and Surgery, KI
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Due to GDPR we are not able to share genomic data, but in case of joined reports anonymized clinical data such as growth parameters or information on malformations will be shared.